CLINICAL TRIAL: NCT04048096
Title: Effects of Krill Oil Supplementation on Muscle Function in Older Adults
Brief Title: Krill Oil and Muscle in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Senior Lecturer in Exercise and Metabolic Health, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200170067
Record Dates: First submitted 2019-07-26; First posted 2019-08-07 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Aging; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 4g/day of mixed vegetable oil supplements
  Interventions: Dietary Supplement: Placebo
- Krill (Experimental): 4g/day krill oil
  Interventions: Dietary Supplement: Krill Oil

INTERVENTIONS:
Dietary Supplement: Krill Oil — Aker Biomarine Superba Krill Oil
  Arms: Krill
Dietary Supplement: Placebo — Mixed vegetable oil
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effects of krill oil supplementation on muscle mass in function in older adults. Half of the participants will receive krill oil supplements and the other half a placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35kg/m2

Exclusion Criteria:

* Diabetes
* severe cardiovascular disease
* seizure disorders
* uncontrolled hypertension (>150/90mmHg at baseline measurement)
* cancer or cancer that has been in remission <5 years
* ambulatory impairments which would limit ability to perform assessments of muscle function
* dementia
* taking medication known to affect muscle (e.g. steroids)
* have an implanted electronic device (e.g. pacemaker/defibrillator/insulin pump)
* on anticoagulant therapy
* allergies to seafood
* regular consumption of more than 2 portions of oily fish per week.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Muscle strength | Change from baseline to 6 months
  knee extensor muscle strength

SECONDARY OUTCOMES:
Change in Grip strength | Change from baseline to 6 months
  Grip strength
Change in Muscle thickness | Change from baseline to 6 months
  Vastus lateralis muscle thickness
Change in Short performance physical battery test | Change from baseline to 6 months
  SPPB
Change in Body Fat | Change from baseline to 6 months
  Measured by BIA
Change in Lean Mass | Change from baseline to 6 months
  Measured by BIA
Change in Fasting glucose | Change from baseline to 6 months
  Fasting glucose
Change in Blood lipids | Change from baseline to 6 months
  Blood lipids
Change in CRP | Change from baseline to 6 months
  CRP
Change in Erythrocyte fatty acid profile | Change from baseline to 6 months
  Erythrocyte fatty acid profile

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Gray, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Stuart Robert Gray, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayman O, Alkhedhairi SA, Combet E, Quinn TJ, Hunter AM, Goodall S, Gray SR. Do the effects of krill oil supplementation on skeletal muscle function and size in older adults differ by sex, age or BMI: A secondary analysis of a randomised controlled trial. J Nutr Health Aging. 2026 Jan;30(1):100747. doi: 10.1016/j.jnha.2025.100747. Epub 2025 Dec 3. PMID 41344001
- [Derived] Alkhedhairi SA, Aba Alkhayl FF, Ismail AD, Rozendaal A, German M, MacLean B, Johnston L, Miller AA, Hunter AM, Macgregor LJ, Combet E, Quinn TJ, Gray SR. The effect of krill oil supplementation on skeletal muscle function and size in older adults: A randomised controlled trial. Clin Nutr. 2022 Jun;41(6):1228-1235. doi: 10.1016/j.clnu.2022.04.007. Epub 2022 Apr 20. PMID 35504165